CLINICAL TRIAL: NCT00625014
Title: Metabolic Effects of Subchronic Dopamine D2 Receptor Blockade by Haloperidol in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Hanno Pijl, Prof dr H Pijl, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P05.009
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Insulin Resistance; Dyslipidemia
Keywords: Insulin resistance; Dyslipidemia; Haloperidol
MeSH Terms: conditions — Insulin Resistance; Dyslipidemias | interventions — Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Healthy men
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Haloperidol — Haloperidol 3 mg/day for 8 days

SUMMARY:
We hypothesized that short-term treatment with haloperidol induces insulin resistance through a mechanistic route that is independent of weight gain. We therefore treated healthy non-obese men with haloperidol for 8 days, and studied the impact of these intervention on glucose and lipid metabolism by hyperinsulinemic euglycemic clamp, isotope dilution technology and indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* 20 kg/m2 < BMI < 26 kg/m2
* Age 20-40 years
* FPG < 6 mmol/L

Exclusion Criteria:

* FPG > 6 mmol/L
* BMI > 26 kg/m2
* Psychiatric disorders and/or use of antipsychotic or antidepressants drugs at present or in the past.
* A positive family history of schizophrenia
* Any significant chronic disease
* Renal, hepatic or endocrine disease
* Use of medication known to influence lipolysis and/or glucose metabolism
* Total cholesterol > 7mmol/L and/or triglycerides > 2 mmol/L
* Recent weight changes or attempts to loose weight (> 3 kg weight gain or loss, within the last 3 months)
* Difficulties to insert an intravenous catheter
* Smoking (current)
* Severe claustrophobia (ventilated hood)
* Recent blood donation (within the last 2 months)
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Extensive sporting activities (more than 10 hours of exercise per week)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To determine the effect of subchronic haloperidol treatment on HGO, whole body peripheral glucose disposal, fatty acid flux and fuel oxidation. | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands